CLINICAL TRIAL: NCT00998569
Title: Neurocognitive Enhancement in Major Depressive Disorder
Acronym: MDDNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Christopher Bowie, Ph.D., Queen's University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PSYC-092-09
Record Dates: First submitted 2009-10-14; First posted 2009-10-20 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurocognitive Enhancement (Experimental): neurocongnitive enhancement
  Interventions: Behavioral: Neurocognitive Enhancement
- Wait List (Other): no intervention
  Interventions: Behavioral: Wait List

INTERVENTIONS:
Behavioral: Neurocognitive Enhancement — Neurocognitive Enhancement Therapy (NET) uses behavioural treatment strategies that are designed to improve a range of cognitive skills. NET uses strategies such as coaching, repetition, practice, teaching, group discussion, and compensation for deficits by using cognitive strengths.
  Arms: Neurocognitive Enhancement
Behavioral: Wait List — Participants will be wait listed for 10 weeks, following which time they will receive the intervention previously described.
  Arms: Wait List

SUMMARY:
The purpose of this study is to examine the effects of neurocognitive enhancement on cognitive abilities and related social and adaptive behaviours in individuals diagnosed with major depressive disorder. Subjects in this study will be randomized to receive Neurocognitive Enhancement Therapy (NET) or to a wait list and then NET . Secondary aims include examining whether the cognitive benefits are potentiated by repeated exposure during in-home practice with complementary exercises. Additionally, the investigators will examine the durability of the effects and their generalization to functional capacity and everyday functional performance after completion of the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female.
2. Subjects will be between the ages of 18 and 65, which is the age range with available normative comparison data.

Exclusion Criteria:

1. Presence of a medical diagnosis that is associated with known cognitive impairments, such as multiple sclerosis, cerebrovascular accident, dementia, or history of traumatic brain injury.
2. Subjects with a reading level below grade 6, as assessed with the Wide Range Achievement Test - Reading Recognition Subtest, will be excluded because of the likelihood of not understanding task instructions.
3. Subjects with uncorrectable vision or hearing impairment that would preclude valid assessments or intervention procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Performance on paper and pencil assessments of neurocognition after treatment, compared to baseline assessment performance | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowie, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada